CLINICAL TRIAL: NCT00885768
Title: Prevalence of Renal Artery Stenosis in Patients Refered for Cardiac Catheterization to Heart Center Hospital in July-September 2008
Brief Title: Prevalence of Renal Artery Stenosis in Patients Referred for Cardiac Catheterization
Acronym: RAS
Status: Completed | Type: Observational
Sponsor: Imam Khomeini Hospital (Other)
Collaborators: Tehran Heart Center (Other)
Responsible Party: Mohammad Reza Khatami, Kidney Research Center
Other Study IDs: RAS001
Record Dates: First submitted 2008-07-11; First posted 2009-04-22 (Estimated); Results first posted 2010-03-23 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2009-04

CONDITIONS: Renal Artery Stenosis
Keywords: RAS(renal Artery Stenosis); Atherosclerosis; angiography
MeSH Terms: conditions — Renal Artery Obstruction; Atherosclerosis | interventions — Cerebral Angiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A: patients with renal artery stenosis
  Interventions: Procedure: angiography

INTERVENTIONS:
Procedure: angiography — all patients undergoing coronary angiography with VISIPAQUE and if they had coronary stenosis then renal artery angiography will be done. the dose of contrast will be chosen according to renal function and clinical conditions which will be varied from 75 to 300 ml.

SUMMARY:
All patients referred for coronary angiography will simultaneously be evaluated for renal artery stenosis and then stenosis more than 50% will be analyzed according to clinical conditions, risk factors and lab data.

DETAILED DESCRIPTION:
Renal Artery Stenosis (RAS) is a common finding in patients with generalized atherosclerosis. It is the cause of 15-20% of end stage renal disease in elderly patients. The prevalence of asymptomatic RAS in general population is unknown but it estimated to be 18% in 7th decade and more than 50% in the 8th. It is critical to find and manage the RAS before it's symptoms appear. The Gold standard for diagnosis of atherosclerotic arterial stenosis is angiography. In this study we will evaluate the prevalence, severity, location and related factors to renal artery stenosis in patients whom referred for coronary angiography in period of July-September in one of the most referral heart center in Iran, "The Tehran heart center" which is doing more than 50 coronary angiography daily.

ELIGIBILITY:
Inclusion Criteria:

* age more than 18 years

Exclusion Criteria:

* contraindication to contrast use
* not signing consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients reffered to the Tehran Heart center for coronary angiography
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2008-07; Primary Completion 2008-09 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Tehran Heart Center, Tehran, Iran

RESULTS

PARTICIPANT FLOW:
Recruitment Details: all patients recruited during 4 months from April 2008 through July 2008 in Tehran Heart Center.
Groups:
- Renal Artery Stenosis: the patients with coronary artery stenosis who have also renal artery stenosis
Period: Overall Study
Arm/Group | Renal Artery Stenosis
Started | 146 (all patients with coronary artery stenosis on angiography entered the study)
Completed | 146 (all patients with including criteria completed the study)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Renal Artery Stenosis
Number analyzed (Participants) | 146
Age Continuous [Mean (Standard Deviation); unit: years] | 61.17 (9.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 95
Region of Enrollment [Number; unit: participants]
  Iran, Islamic Republic of | 146
the adult patients with coronary artry disease [Number; unit: participants] — when the reffered patients for coronary angiography have been proved to have significant coronary artery stenosis then the angiography of renal artery were performed.
  participants
    <=18 years | 0
    Between 18 and 65 years | 127
    >=65 years | 19
the patients with coronary artery disease [Number; unit: participants] | 146

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Renal Artery Stenosis (RAS)
Time Frame: 2 months
Reporting Status: Not Posted

2. Primary Outcome: The Number of Patients With Renal Artery Stenosis
Description: the prevalence of renal artery stenosis in patients with coronary artery disease
Time Frame: 3months
Measure: Number; unit: participants
Arm/Group | Renal Artery Stenosis
Number analyzed (Participants) | 146
participants | 146

ADVERSE EVENTS:
Arm/Group | Renal Artery Stenosis
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes